CLINICAL TRIAL: NCT03676114
Title: Effect of Perioperative Low Dose Ketamine on Postoperative Recovery in Patients Undergoing Breast Cancer Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Han Yuan (Other)
Responsible Party: Sponsor-Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XuzhouMedSch3
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Ketamine; Breast Cancer Surgery; Postoperative Recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Experimental)
  Interventions: Drug: ketamine
- normal saline group (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: ketamine — 0.5mg/kg intravenous ketamine injection before incision followed by 0.25mg/kg/hr intravenous ketamine infusion during the operation
  Arms: ketamine group
Drug: Normal saline — Same volume of normal saline will be administrated
  Arms: normal saline group

SUMMARY:
Breast cancer patients often have perioperative emotional disorders such as anxiety and depression, which can lead to poor quality of recovery.This study aims to determine whether ketamine could improve the quality of recovery in breast cancer patients. Meanwhile, it will show if ketamine could improve anxiety, depression, postoperative pain and fatigue.This trial also will bring great concerns on patients' mental health perioperatively and explore the measures to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists Grade I-II
2. Patients undergoing elective breast cancer surgery under general anesthesia

Exclusion Criteria:

1. Unstable hypertension, history of heart disease
2. Hepatic or renal dysfunction
3. Patients undergoing chemotherapy before surgery
4. Have a history of chronic pain or chronic use of analgesic
5. Have mental illness or can't cooperate with investigators
6. Have a history of ketamine allergy

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
QoR40 score | the first day after surgery
  Quality of recovery will be evaluated by Quality of Recovery 40 (QoR40),which assesses five dimensions of recovery (physical comfort,emotional state, physical independence , physiological support and pain ). Each item is rated on a five-point Likert scale: none of the time, some of the time, usually, most of the time, and all the time. The total score on the QoR40 ranges from 40 (poorest quality of recovery) to 200 (best quality of recovery).

SECONDARY OUTCOMES:
ICFS scores | Postoperative 3 days, 7 days and 30 days
  Fatigue state will be evaluated by Identity Consequence Fatigue Scale (ICFS).ICFS is based on a score of 31-173, higher scores representing worse state of fatigue.
HADS scores | Postoperative 2 days and 3months
  Perioperative emotion will be evaluated by the hospital anxiety and depression scale（HADS）.The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Chronic Pain | 3 months after surgery
  The incidence of chronic pain at 3 months after surgery
NRS pain scores | at 4 hours, 24 hours, and 48 hours after surgery
  Evaluate the severity using numerical rating scale（NRS）, where zero mean no pain and 10 the worst imaginable pain.
Postoperative complications | Postoperative 1 day, 2 days and 3 days
  hallucination, nightmare and delirium will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China